CLINICAL TRIAL: NCT00564577
Title: Dose-Finding Study of WS6788A and LSN03-016011/A Enterotoxigenic E. Coli (ETEC) Challenge Strains That Express CS17
Brief Title: Dose-Finding Study of WS6788A and LSN03-016011/A Enterotoxigenic E. Coli ETEC Challenge Strains That Express CS17
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: Naval Medical Research Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: CIR 193 (B)
Record Dates: First submitted 2007-11-26; First posted 2007-11-28 (Estimated); Last update posted 2017-04-11 (Actual); Status verified 2017-04

CONDITIONS: Travelers' Diarrhea
Keywords: Diarrhea ETEC

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CFA/I and CS17 challenge strain (Other): Colonization factor antigen (CFA/I) and CS17 challenge strainAscending dose finding study in 5-10 subjects per dose; to identify the dose able to give a diarrheal attack rate greater than or equal to 80%.
  Interventions: Biological: CFA/I and CS17 challenge strain

INTERVENTIONS:
Biological: CFA/I and CS17 challenge strain — Wild type ETEC strain expressing the colonization factor CS17, and heat labile (LT) enterotoxin
  Other Names: Experimental

SUMMARY:
This will be a strain and dose-finding study in which LSN03-016011/A ETEC will be administered at a starting inoculum of 5x108 cfu to 5 subjects to establish a human disease model. If 80% attack rate (AR) is achieved without high output diarrhea, the same inoculum will be given to 10 more subjects for confirmation of AR. If 80% AR is not achieved, attack rate and severity of disease will be evaluated to determine if the dose should be increased. The same sequence may be conducted with WS6788A if applicable. If the LSN strain causes high output diarrhea the dose will be adjusted down and further dose characterization continued. An iterative process will be used to select the optimal strain and dose with each step reviewed and approved by the medical monitor.

DETAILED DESCRIPTION:
This is a phase 1, open-label, strain and dose-finding study designed to establish a human challenge model for CS17+ ETEC that causes > 80% attack rate without causing high output diarrhea. Based on the strain histories, testing will commence using LSN03-016011/A. This strain was isolated from a naïve adult U.S. citizen living in Turkey with a typical clinical presentation for ETEC diarrheal disease and no bacterial co-pathogens isolated from the stool. The host is representative of the study population for this study and for future efficacy studies with anti-CS17+ ETEC vaccines. As shown in the figure below, 5x108 cfu of ETEC strain (LSN03-016011/A) will initially be administered to 5 subjects. If an attack rate of >80% (at least 4/5 subjects) occurs with no high output diarrhea, results will be confirmed in an additional 10 subjects. Additionally, an inoculum at least ½ log lower (1x108) (depending on the severity of illness documented) may be administered to 10 subjects to characterize the dose-response relationship. If the 5x108 cfu inoculum does cause high output diarrhea, then the inoculum will be reduced appropriatelyIf the 5x108 cfu of LSN03-016011/A does not cause a > 80% attack rate, the next step will depend on the observed attack rate and severity of illness. A low attack rate with mild disease would prompt a change to the alternate strain (WS7688A) for testing, using the same pathway used with the LSN strain . An attack rate < 80% with most diarrhea classified as at least moderate diarrhea would prompt an upward adjustment of the LSN inoculum appropriate to the findings. The decision to move up or down in inoculum or to change CS17 + strains will only occur with the concurrence of the medical monitor. Following each step in the strain and dose finding iterations, a report summarizing the results of that step, and detailing the planned next step will be signed by the principal investigator and the medical monitor. The maximum dose of either strain is 1 X 109. The anticipated maximum number of subjects planned for this study is 25.

Subjects will be admitted to the inpatient facility on study day -1. On study day 0, subjects will have their morning meal, fast for 90 minutes, and then be given 120mL of sodium bicarbonate buffer to neutralize stomach acidity. Approximately one minute later they will ingest the appropriate dose and strain (either LSN03-016011/A or WS6788A ) of CS17+ ETEC diluted in 30mL sodium bicarbonate buffer. Doses of the challenge inoculum will be prepared by one of the study staff microbiologists. Treatment with antibiotics will start on study day 5, or earlier if criteria for early antibiotic treatment are fulfilled. Subjects will be discharged when they feel well and have 2 consecutive stool cultures negative for CS17+ ETEC.

For each group of 5 study subjects, the study period will include the screening period, one month for the inpatient and outpatient phases, and six-months for the final phone check. The study period, accounting for the serial scheduling of multiple groups of 5, processing immunology specimens, study analysis and report writing, is 1 ½ years.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female between 18 and 45 years of age, inclusive.
2. General good health, without significant medical illness, abnormal physical examination findings or clinical laboratory abnormalities as determined by principal investigator or principal investigator in consultation with the medical monitor and sponsor.
3. Demonstrate comprehension of the protocol procedures and knowledge of ETEC illness by passing a written examination (pass grade ≥ 70%)
4. Willing to participate after informed consent obtained.
5. Available for all planned follow-up visits.
6. Negative serum pregnancy test at screening and a negative urine pregnancy test on the day of admittance to the inpatient phase for female subjects of childbearing potential. Females of childbearing potential must agree to use an efficacious hormonal or barrier method of birth control during the study. Abstinence is acceptable. Female subjects unable to bear children must have this documented (e.g., tubal ligation or hysterectomy).

Exclusion Criteria:

1. Presence of a significant medical condition, (e.g. psychiatric conditions or gastrointestinal disease, such as peptic ulcer, symptoms or evidence of active gastritis or gastroesophageal reflux disease, inflammatory bowel disease, alcohol or illicit drug abuse/dependency), or other laboratory abnormalities which in the opinion of the investigator precludes participation in the study.
2. Immunosuppressive illness or immunoglobulin A (IgA) deficiency (below the normal limits)
3. Positive serology results for HIV, HBsAg, or Hepatitis C virus (HCV) antibodies.
4. Significant abnormalities in screening lab hematology, serum chemistry, urinalysis or EKG (EKG in subjects ≥ 40 years), as determined by PI or PI in consultation with the medical monitor and sponsor.
5. Allergy to fluoroquinolones, trimethoprim-sulfamethoxazole, or ampicillin/penicillin (excluded if allergic to two of three).
6. Fewer than 3 stools per week or more than 3 stools per day as the usual frequency, loose or liquid stools other than on an occasional basis.
7. History of diarrhea in the 2 weeks prior to planned inpatient phase
8. Regular use of laxatives or any agent that increase gastric pH (regular defined as at least weekly).
9. Use of antibiotics during the 7 days before bacterial dosing or proton pump inhibitors, H2 blockers, or antacids within 48 hours of dosing.
10. Travel to countries where ETEC or cholera infection is endemic (most of the developing world) within two years prior to dosing.
11. History of vaccination for or ingestion of ETEC, cholera, or LT toxin.
12. Stool culture (collected no more than 1 week prior to admission) positive for CS17 + ETEC or other bacterial enteric pathogens (Salmonella, Shigella and Campylobacter).
13. Use of any investigational product within 30 days preceding the receipt of the challenge inoculum, or planned use during the active study period.
14. Use of any medication known to affect the immune function (e.g., corticosteroids and others) within 30 days preceding receipt of the challenge inoculum or planned use during the active study period.

Ages: 15 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 13 (Actual)
Dates: Start 2006-09 (Actual); Primary Completion 2007-06-13 (Actual); Study Completion 2007-06-13 (Actual)

PRIMARY OUTCOMES:
Development of diarrhea | 120 hours after challenge

SECONDARY OUTCOMES:
Development of moderate to severe diarrhea | 120 hours after challenge

CONTACTS AND LOCATIONS:
Overall Officials: Robin McKenzie, M.D., Principal Investigator — Johns Hopkins Bloomberg School of Public Health
Locations (2):
- United States (2):
  - Center for Immunization Research - Johns Hopkins Bloomberg School of Public Health, Baltimore, Maryland
  - General Clinical Research Center of the Johns Hopkins Hospital, Baltimore, Maryland

IPD SHARING:
Plan to Share IPD: No